CLINICAL TRIAL: NCT04211116
Title: Central Venous Catheters in Pediatric Anesthesia and Intensive Care: Prospective Observational Trial
Brief Title: Central Venous Catheters in Pediatric Anesthesia and Intensive Care
Acronym: PEDCVC
Status: Completed | Type: Observational
Sponsor: Brno University Hospital (Other)
Responsible Party: Principal Investigator, Petr Štourač, MD, assoc.prof.MD,Ph.D, Brno University Hospital
Other Study IDs: KDAR FN Brno 2020/1
Record Dates: First submitted 2019-12-22; First posted 2019-12-26 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Central Line
Keywords: Central line; Pediatric patient; Insertion; Cannulation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pediatric patients indicated to CVC insertion: Paediatric patients indicated to central venous line insertion
  Interventions: Device: Central venous line insertion

INTERVENTIONS:
Device: Central venous line insertion — Pediatric patients indicated to central venous line insertion
  Other Names: Central venous line cannulation

SUMMARY:
Securing the intravenous line is one of the fundamental interventions in paediatric anaesthesia and intensive care. Central venous catheters (CVC) are indicated for long-term stay in intensive care unit (ICU), in case of circulatory instability and the need for vasopressor therapy, for hypertonic solutions administration and parenteral nutrition. The dominant method of CVC insertions is the Seldingers´ method (over the wire) and ultrasound real-time navigation in recommended. Ultrasound-guided (USG) CVC insertion however requires experience personnel and relevant training.This could be the main reason, that CVC the real-time ultrasound navigation is still not adequately implemented into the clinical practice.

DETAILED DESCRIPTION:
After Ethics committee approval, patients indicated for CVC insertions will be included. Based on the observational design of the trial, the method of insertion (Real-time ultrasound navigation versus anatomical-based CVC insertion) will be based on operators´ decision.The indication for CVC insertion, primary planned site of insertion, USG implementation, site of actual CVC cannulation and associated complications will be recorded. The primary aim of the study was to compare the effectivity of Real-time ultrasound navigation versus anatomical-based CVC insertion in paediatric patients and the 1st percutaneous puncture success rate. The secondary aims will be the incidence of associated complications and the time form first percutaneous puncture, to definitely securing the CVC in place. The primary hypothesis is that the Ultrasound-guided CVC insertion is superior, with the higher overall success, higher first attempt success rate and with lower incidence of associated complications.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients within the age limit indicated for CVC insertion

Exclusion Criteria:

* Outside the age limit

Max Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric patients
Sampling Method: Non-Probability Sample
Enrollment: 107 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-02-15 (Actual)

PRIMARY OUTCOMES:
Overall success and first attempt success rate | During CVC insertion
  The overall success rate and first attempt success rate will be evaluated between ultrasound-guided and anatomical-based navigation

SECONDARY OUTCOMES:
Incidence of complications | 24 hours from CVC insertion
  Incidence of arterial puncture, hemothorax and/or pneumothorax incidence, incidence of CVC malposition will be recorded
Time of insertion | During CVC insertion
  The time from first percutaneous puncture to CVC insertion will be monitored and evaluated between

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Brno, Brno, State, Czechia

IPD SHARING:
Plan to Share IPD: Undecided